CLINICAL TRIAL: NCT05084339
Title: Glucose Homeostasis, Metabolomics and Pregnancy Outcomes After Bariatric Surgery
Acronym: GLORIA
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Antwerp (Other); University Hospital, Ghent (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Onze Lieve Vrouw Hospital (Other); Imelda Hospital, Bonheiden (Other); AZ Sint-Lucas Brugge (Other); General Hospital Groeninge (Other)
Responsible Party: Sponsor
Other Study IDs: S65734
Record Dates: First submitted 2021-09-20; First posted 2021-10-19 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Bariatric Surgery Status Complicating Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant group with bariatric surgery: pregnant women with a history of gastric bypass or sleeve gastrectomy
  Interventions: Diagnostic Test: CGM
- matched pregnant group without history of bariatric surgery: age-and BMI matched pregnant women without history of bariatric surgery
  Interventions: Diagnostic Test: CGM

INTERVENTIONS:
Diagnostic Test: CGM — blinded CGM used at 4 different time points in pregnancy

SUMMARY:
The aim of the GLORIA study is to determine whether an altered glucose metabolism (with more hypoglycaemia and glycaemic variability) and altered metabolomics during pregnancy after bariatric surgery contribute to the increased risk for adverse pregnancy outcomes such as small-for-gestational age infants. In addition, the investigators also aim to evaluate whether continuous glucose monitoring (CGM) can be used to diagnose gestational diabetes (GDM).

DETAILED DESCRIPTION:
The GLORIA study is a Belgian multicenter prospective cohort study. The investigators aim to recruit 95 pregnant women after bariatric surgery (gastric bypass or sleeve gastrectomy) and as a control group, an age and BMI-matched cohort of 95 pregnant women without bariatric surgery. Participants will be recruited before 12 weeks of pregnancy. To evaluate glucose homeostasis, a masked CGM will be used for 10 days during each trimester in pregnancy and at the time of screening for GDM (at 24-28 weeks). The primary outcome is the mean glycaemia levels and glycaemic variability (SD) measured by CGM in pregnancy. At the different time points, anthropometric measurements (including body composition), food diary, questionnaires and micronutrients will be evaluated. In addition, in collaboration with the lab of Cristina Legido Quigle from the Steno Diabetes Center in Copenhagen, metabolomics will be analyzed. Women with a history of bariatric surgery will receive screening for GDM between 24-28 weeks of pregnancy by performing self- monitoring of blood glucose (SMBG) with a glucometer during one week. In addition to SMBG, women will receive a masked CGM during one week.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years and with a singleton pregnancy with ultrasound-confirmed gestational age up to 11 weeks and 6 days
* for the group with bariatric surgery: history of gastric bypass (RYBG) or sleeve gastrectomy (SG)
* Participants need to speak and understand Flemish, French or English and have e-mail access.

Exclusion Criteria:

* multiple pregnancy
* pregnancy ≥12 weeks
* other types of bariatric surgery than RYBG or SG
* known pregestational diabetes
* a physical or psychological disease likely to interfere with the conduct of the study
* medications known to interfere with glucose metabolism.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 95 pregnant women with a history of bariatric surgery (RYBG or SG) and 95 age-and BMO matched pregnant women without history of bariatric surgery
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
mean glycaemia | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  mean glycaemia measured by CGM
Standard deviation of glycaemia | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  SD measured by CGM

SECONDARY OUTCOMES:
time <54mg/dl | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  time <54mg/dl measured by CGM
glycaemic variability measured by coefficient of variation (CV) | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  CV measured by CGM
glycaemic variability measured by mean amplitude of glucose excursions (MAGE) | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  MAGE measured by CGM
time <70mg/dl | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  time <70mg/dl measured by CGM
time <63mg/dl | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  time <63mg/dl measured by CGM
time <50mg/dl | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  time <50mg/dl measured by CGM
low blood glucose index (LBGI) | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  low blood glucose index (LBGI) based on CGM
time > 120mg/dl | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  time >120mg/dl measured by CGM
time > 140mg/dl | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  time >140mg/dl measured by CGM
time > 180mg/dl | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  time >180mg/dl measured by CGM
prevalence of gestational diabetes | 24-28 weeks of pregnancy
  gestational diabetes based on capillairy monitoring or oral glucose tolerance test
gestational weight gain | at end of pregnancy
  total gestational weight gain in pregnancy
preterm delivery | delivery
  delivery <37 weeks of pregnancy
cesarean sections | delivery
  planned and emergency cesarean sections combined
large-for-gestational age infant | delivery
  gestational age adjusted birth weight >90th percentile according to the standardized Flemish birth charts adjusted for parity and sex
small-for-gestational infant | delivery
  gestational age adjusted birth weight <10th percentile according to the standardized Flemish birth charts adjusted for parity and sex
neonatal hypoglycaemia | delivery
  neonatal hypoglycaemia requiring intravenous dextrose
Neonatal intensive care admission (NICU) | delivery
  NICU admission defined as requiring a duration of at least 24 h
gestational hypertension | delivery
  gestational hypertension ≥20 weeks of gestation: blood pressure ≥140/90mmHg
pre-eclampsia | delivery
  pre-eclampsia [≥20 weeks of gestation: new onset of hypertension and proteinuria or the new onset of hypertension and significant end-organ dysfunction with or without proteinuria (dipstick ≥ 2+, ≥0.3 g protein/24 hours or ≥30 mg/dL protein in spot urine or spot urine protein / creatinine ratio ≥30 mg protein/mmol creatinine)
micronutrient deficiencies | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy and 30-34 weeks of pregnancy
  vitamin A, vitamin D, B12, folate, prothrombin time and iron
body fat percentage women | between 6-12 weeks of pregnancy
  body fat measured by bioelectrical impedance analysis
body fat percentage newborns | within 3 days after birth
  body fat calculated by measurements of skinfolds at triceps, flank and subscapular
fetal abdominal circumference (AC) | at 12, 20, 30 and 34 weeks of gestation
  fetal abdominal circumference (AC) to evaluate fetal body composition
fetal abdominal subcutaneous fat thickness (ASCF) | at 12, 20, 30 and 34 weeks of gestation
  fetal abdominal subcutaneous fat thickness (ASCF) to evaluate fetal body composition
placental function | at 12, 20, 30 and 34 weeks of gestation
  the pulsatility index (PI) of the Doppler wave in the arteriae uterinae at 12 weeks and in the arteria umbilicalis at 20, 30 and 34 weeks of gestation.
macronutrient intake baseline | between 6-12 weeks of pregnancy
  food diary taken in early pregnancy
macronutrient intake in pregnancy | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  frequency food questionnaire
physical activity | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  the Kaiser physical activity survey
symptoms of depression | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  the 20-item Center for Epidemiologic Studies-Depression (CES-D) questionnaire
symptoms of anxiety | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  six-item short-form the State-Trait Anxiety Inventory (STAI) questionnaire on anxiety
index of quality of life | between 6-12 weeks of pregnancy, 18-22 weeks of pregnancy, 24-28 weeks of pregnancy and 30-34 weeks of pregnancy
  36-Item Short Form Health Survey (SF-36) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Benhalima, MD PhD, Principal Investigator — UZ Leuven
Locations (8):
- Belgium (8):
  - OLV-Aalst-Asse, Aalst
  - UZA, Antwerp
  - ZNA Antwerpen, Antwerp
  - Imelda Bonheiden, Bonheiden
  - AZ St-Jan Brugge, Bruges
  - UZ Gent, Ghent
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deleus E, Bochanen N, Ceulemans D, Debunne H, Denys B, Devlieger R, Geerts I, Laenen A, Jochems L, Lannoey E, Lannoo M, Loccufier A, Maes T, Marlier J, Morrens A, Myngheer N, Tierens L, Vandenberghe G, Van den Bruel A, Van den Haute L, Van der Schueren B, Van Pottelbergh I, Benhalima K. Glucose Homeostasis, Metabolomics, and Pregnancy Outcomes After Bariatric Surgery (GLORIA): Protocol for a Multicentre Prospective Cohort Study. J Clin Med. 2025 Jul 7;14(13):4782. doi: 10.3390/jcm14134782. PMID 40649156